CLINICAL TRIAL: NCT03007511
Title: Safety and Usability Evaluation of the Fidmi Low-Profile Enteral Feeding Device
Acronym: Fidmi
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to limited financial resource
Sponsor: Fidmi Medical (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Fidmi
Record Dates: First submitted 2016-12-21; First posted 2017-01-02 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Feeding Tube; Dysphagia
Keywords: Percutaneous Endoscopic Gastrostomy; Feeding tube; Enteral nutrition; Endoscopy; Gastrointestinal
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fidmi (Experimental): Placement of Fidmi enhanced enteral feeding device; internal tubes replacement during follow up and device removal after 3 month from placement Fidmi enhanced enteral feeding device
  Interventions: Device: Fidmi enhanced enteral feeding device

INTERVENTIONS:
Device: Fidmi enhanced enteral feeding device — Fidmi enhanced enteral feeding device is intended to provide nutrition to a patient directly into the stomach through a stoma. The Fidmi PEG device would be investigated in this study on patients suffering from dysphagia, who are scheduled for PEG procedure in order to improve surgical initial insertion, device replacement and removal.
  Other Names: Low profile Gastrostomy; Percutaneous Endoscopic Gastrostomy (PEG) device

SUMMARY:
A First In Human Usability Open Label trial will be performed using the Fidmi Feeding device on 20 adult patients with a need for enteral feeding. The primary outcome will be to evaluate safety, usability and discomfort throughout the study

DETAILED DESCRIPTION:
A gastrostomy is a feeding tube that communicates from the skin directly into the stomach. It is a device frequently used in patients that have feeding difficulties or are unable to maintain normal growth via oral feeds.

Currently there are many solutions in the market for long-term enteral feeding, however none of them provide comfort and autonomy to their users, since they have a high probability of dislodgement, clogging, leakage and are bulky.

The Fidmi Medical PEG Feeding Tube and Accessories are to provides food, liquids and medications into the stomach of patients who are having difficulty of swallowing. Fidmi Feeding Device is the first presented "low-profile device from day 1", easily hidden under clothing and not limiting mobility. Unlike other solutions, Fidmi device is resistant to dislodgement due to a semi-rigid internal bumper, and avoids clogging thanks to a disposable insert to deliver the nutrition.

Fidmi device consists of 1) a rigid-core silicone bumper that prevents dislodgment, 2) a disposable internal tube replacement for a daily nutrition supply and prolonged patency, and 3) an external flexible bolster that keeps the stoma site ventilated and stable. The disposable insert is placed inside the feeding port and is replaced every 1-2 weeks to avoid clogging, extend the product life, and improve the cleanliness and hygiene of the tube. Disposable tube replacement is easy and safe and can be done by the patients themselves or their caregivers as the tract is never compromised and there is no need for a physician verification. The device is eventually removed in a simple procedure that can be done by the caregiver or patient themselves. Fidmi device obtain a tool that dismantles the internal bumper into small parts that are naturally expelled from the body for trauma free-removal.

The Fidmi Feeding device would be inserted into eligible enrolled patients who would be followed up during a period of 3 months until device removal. Safety, usability and discomfort parameters would be monitored following 2, 30, 60, 90 and 120 days following the insertion procedure.

In case a new Fidmi PEG device is requested by a patient: additional duration of 120 days±14 days will be added.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient 18 up to 90 years.
2. Consecutive adult patients suffering from dysphagia with need for enteral feeding (PEG).
3. Ability to give informed consent for the study by patient or legal guardian.
4. Willingness to undergo 4 follow up visits 1, 3 and 4 months following PEG insertion/replacement, as well as unscheduled sick visits.

Exclusion Criteria:

1. Pregnancy (all women of child-bearing age would be questioned and told by the consenting physician regarding that criteria).
2. All current practice PEG contraindication
3. Acute gastrointestinal bleeding
4. Extreme obesity patients (BMI>40)
5. Emergency endoscopy
6. Infectious disease local or systemic (e.g.- sepsis, pancreatitis)
7. Known esophageal pathology (e.g.- stenosis, eosinophilic esophagitis, varices, achalasia)
8. In case of PEG replacement: lack of a well healed gastrostomy or Infection around the insertion site.
9. Known gastric pathology that may prevent safe device insertion, feeding, removal and Bumper flanges expulsion according to the investigator discretion.
10. Any history of bowel obstruction, pseudo-obstruction.
11. Crohn's disease
12. Recurrent vomiting
13. Inability to tolerate sedated upper endoscopy due to cardio-pulmonary instability or other contraindication to endoscopy
14. Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment related Adverse Events | Through study completion, an average of 4 months
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Ease of the device placement procedure (using the 10-point Visual analogue scale satisfaction) | at Day 0
  Scored by the investigator performing the procedure
Ease of the device removal procedure (using the 10-point Visual analogue scale satisfaction) | at 3 Months
  Scored by the investigator performing the procedure
Accidental dislodgements | until device removal at 3 months
  Number of accidental dislodgements during study follow up
Patient Pain | at 3 months
  Patient Pain on the Visual Analog Scale during device removal and sedative medication if administrated

OTHER OUTCOMES:
Validate (True/False) correct (color) selection of 'Measuring Cannula' by residual tube measurement | at day 0
  design outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Harold, MD, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem, Ein Kerem
  - Shaare Zedek Medical Center, Jerusalem

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT03007511/Prot_000.pdf